CLINICAL TRIAL: NCT00300053
Title: A DB, Randomized, Placebo-controlled Study of the Tolerability, Efficacy, Safety, and Dose Range of Intramyocardial CLBS14 for Reduction of Angina Episodes in Patients With Refractory Chronic Myocardial Ischemia (ACT34-CMI)
Brief Title: ACT34-CMI -- Adult Autologous CD34+ Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24779
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Myocardial Ischemia
Keywords: angina
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CLBS14: Low-Dose Group (Experimental): 10 intramyocardial injections of 0.2 mL each of auto-CD34+ cells at a dose of 1 x 10^5 (=100000) cells/kg bodyweight
  Interventions: Biological: CLBS14 (low-dose)
- CLBS14: High-Dose Group (Experimental): 10 intramyocardial injections of 0.2 mL each of auto-CD34+ cells at a dose of 5 x 10^5 (=500000) cells/kg bodyweight
  Interventions: Biological: CLBS14 (high-dose)
- Placebo injection (Placebo Comparator): 10 intramyocardial injections of 0.2 mL each of 0.9% NaCl (saline) in 5% autologous plasma
  Interventions: Biological: placebo injection

INTERVENTIONS:
Biological: CLBS14 (low-dose) — Eligible subjects will receive subcutaneous injections of 5 µg/kg/day G-CSF for 5 days to mobilize CD34+ cells from the bone marrow to the peripheral blood. Mononuclear cells (MNCs) will be collected via apheresis on day 5. On the day of the cell/placebo injection (day 6), the apheresis product will be enriched for CD34+ cells using the Isolex 300i Magnetic Cell Selection System (Baxter Healthcare). Autologous CD34+ cells will be delivered in 10 intramyocardial injections of 0.2 mL at a dose of 1 x 10^5 (=100000) cells/kg bodyweight each using the MyoStar injection catheter (Biosense Webster, Inc.) into the target areas of myocardial ischemia.
  Other Names: G-CSF mobilized, autologous CD34+ cells
  Arms: CLBS14: Low-Dose Group
Biological: CLBS14 (high-dose) — Eligible subjects will receive subcutaneous injections of 5 µg/kg/day G-CSF for 5 days to mobilize CD34+cells from the bone marrow to the peripheral blood. Mononuclear cells (MNCs) will be collected via apheresis on day 5. On the day of the cell/placebo injection (day 6), the apheresis product will be enriched for CD34+ cells using the Isolex 300i Magnetic Cell Selection System (Baxter Healthcare). Autologous CD34+ cells will be delivered in 10 intramyocardial injections of 0.2 mL at a dose of 5 x 10^5 (=500000) cells/kg bodyweight each using the MyoStar injection catheter (Biosense Webster, Inc.) into the target areas of myocardial ischemia.
  Other Names: G-CSF mobilized, autologous CD34+ cells
  Arms: CLBS14: High-Dose Group
Biological: placebo injection — Eligible subjects will receive subcutaneous injections of 5 µg/kg/day G-CSF for 5 days to mobilize CD34+ cells from the bone marrow to the peripheral blood. Mononuclear cells (MNCs) will be collected via apheresis on day 5. On the day of the cell/placebo injection (day 6), the apheresis product will be enriched for CD34+ cells using the Isolex 300i Magnetic Cell Selection System (Baxter Healthcare). Placebo will be delivered in 10 intramyocardial injections of 0.2 mL each of 0.9% NaCl (saline) in 5% autologous plasma into the target areas of myocardial ischemia.
  Other Names: 0.9% NaCl (saline) in 5% autologous plasma
  Arms: Placebo injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intramyocardial injections of CLBS14 in patients with refractory chronic myocardial ischemia.

DETAILED DESCRIPTION:
This is a double-blind, prospective, randomized, placebo-controlled trial to determine the tolerability, efficacy, safety and dose range of intramyocardial injections of adult autologous CD34+ cells mobilized with granulocyte colony stimulating factor (G-CSF) for the reduction of angina episodes in patients with refractory chronic myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Canadian Cardiovascular Society (CCS) functional class III or IV chronic refractory angina
* subjects without control of their angina symptoms, in spite of maximal tolerated doses of anti-anginal drugs, must be on optimal therapy for their angina and on a stable anti-anginal medication regimen for at least 1 month prior to entering the screening period of the study
* identified as unsuitable for conventional revascularization
* recent coronary angiogram (within the last 12 months) to document the coronary anatomy and to verify the revascularization procedures
* subjects must have objective evidence of inducible ischemia or viable myocardium in the potential target injection zone
* a left ventricular ejection fraction equal to or greater than 25% by ECHO or single photon emission computed tomography (SPECT) at screening
* subjects must experience at minimum an average of 7 angina or anginal equivalent episodes per week
* subjects must be able to complete a minimum of 3 minutes but nor more than 10 minutes on a treadmill following the Modified Bruce Protocol
* subjects must experience angina or anginal equivalent episodes during the screening exercise treadmill test
* female subjects must either be no longer capable of reproduction or using medically valid contraception to prevent pregnancy during the study
* subjects must be willing and able to comply with specified follow-up evaluations

Exclusion Criteria:

* predominant congestive heart failure
* myocardial infarction within 60 days of treatment
* successful or partially successful coronary revascularization procedures (any vessel) within 6 months of study enrollment
* placement of a bi-ventricular pacemaker for cardiac resynchronization therapy (CRT) for heart failure in the past 90 days
* documented stroke or transient ischemic attack (TIA) within 60 days of study enrollment
* history of moderate to severe aortic stenosis or severe aortic insufficiency; severe mitral stenosis or severe mitral insufficiency
* prosthetic aortic valve replacement
* evidence of any life-threatening arrhythmia that requires intervention on the 24-hour Holter monitor. Life-threatening arrhythmia that is successfully treated with an implantable cardioverter defibrillator (ICD) is not exclusionary.
* splenomegaly and/or severe co-morbidity associated with a reduction in life expectancy of less than 1 year, such as chronic medical illness (ie, severe chronic obstructive pulmonary disease, renal failure or cancer [exceptions: in-situ skin cancer or fully removed skin cancer other than melanoma, in-situ cervical cancer, or cancer free for 5 years with no history of a stem cell transplant])
* sickle cell disease or sickle cell trait
* platelet count greater than 10% above the upper limit of normal or a platelet count below 100,000 if on Clopidogrel or 50,000 without Clopidogrel
* hematocrit <30%
* serum creatinine >2.5 mg/dL
* any clinically significant laboratory abnormality on screening laboratories
* currently enrolled in another IDE or IND that has not completed the protocol required primary follow-up period (excludes 15 year follow up of gene therapy trials)
* history of alcohol or drug abuse within 3 months of screening
* joint or peripheral vascular disease or neurologic disease that severely limits treadmill walking
* chronic obstructive pulmonary disease that severely limits walking or FEV1 <30% predicted
* females who are pregnant or lactating
* female subjects who are capable of reproduction and will not use medically valid contraception to prevent pregnancy during the study
* subjects who test positive for HIV, hepatitis B or hepatitis C, or are on chronic immunosuppressive medications or have had a prior stem cell transplant
* subjects with a known hypersensitivity to E. coli-derived proteins, or to any component of Neupogen (Filgrastim) or G-CSF
* subjects who have a significant psychiatric disorder or mental disability that could interfere with the subject´s ability to provide informed consent and/or comply with protocol procedures

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caladrius Study DIrector, Study Director — Lisata Therapeutics, Inc.
Locations (26):
- United States (26):
  - Cardiology PC, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Scripps Memorial Hospital, La Jolla, California
  - Stanford University Hospital and Clinics, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Central Florida Cardiology Group, Orlando, Florida
  - Saint Joseph's Research Institute, Atlanta, Georgia
  - Northwestern University Medical Center, Bluhm Cardiovascluar Institute, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinic, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Caritas Saint Elizabeth's Medical Center, Boston, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical College of Cornell University, New York, New York
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Swedish Heart & Vascular - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Medical School, Madison, Wisconsin
  - Comprehensive Cardiovascular Care Group, Milwaukee, Wisconsin

REFERENCES:
- [Result] Losordo DW, Henry TD, Davidson C, Sup Lee J, Costa MA, Bass T, Mendelsohn F, Fortuin FD, Pepine CJ, Traverse JH, Amrani D, Ewenstein BM, Riedel N, Story K, Barker K, Povsic TJ, Harrington RA, Schatz RA; ACT34-CMI Investigators. Intramyocardial, autologous CD34+ cell therapy for refractory angina. Circ Res. 2011 Aug 5;109(4):428-36. doi: 10.1161/CIRCRESAHA.111.245993. Epub 2011 Jul 7. PMID 21737787
- [Result] Henry TD, Schaer GL, Traverse JH, Povsic TJ, Davidson C, Lee JS, Costa MA, Bass T, Mendelsohn F, Fortuin FD, Pepine CJ, Patel AN, Riedel N, Junge C, Hunt A, Kereiakes DJ, White C, Harrington RA, Schatz RA, Losordo DW; ACT. Autologous CD34+ Cell Therapy for Refractory Angina: 2-Year Outcomes From the ACT34-CMI Study. Cell Transplant. 2016;25(9):1701-1711. doi: 10.3727/096368916X691484. Epub 2016 May 4. PMID 27151378
- [Derived] Povsic TJ, Losordo DW, Story K, Junge CE, Schatz RA, Harrington RA, Henry TD. Incidence and clinical significance of cardiac biomarker elevation during stem cell mobilization, apheresis, and intramyocardial delivery: an analysis from ACT34-CMI. Am Heart J. 2012 Nov;164(5):689-697.e3. doi: 10.1016/j.ahj.2012.06.022. PMID 23137499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 26 clinical sites in the US.
Pre-assignment Details: Of 321 enrolled subjects, 147 were screen failures. Of 174 subjects who started cell mobilization, 1 did not complete the mobilization due to possible left ventricular mural thrombosis. Of 173 subjects who completed mobilization, 168 were randomized to 1 of 3 treatment groups, of which 1 was discontinued prior to treatment due to coagulopathy.
Groups:
- CLBS14: Low-Dose Group: Intramyocardial injections of auto-CD34+ cells at low dose (1 x 10^5 cells/kg bodyweight)
- CLBS14: High-Dose Group: Intramyocardial injections of auto-CD34+ cells at high dose (5 x 10^5 cells/kg bodyweight)
- Placebo Control: Intramyocardial placebo injections
Period: Overall Study
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control
Started | 55 (started = randomized and treated/injected) | 56 (started = randomized and treated/injected) | 56 (started = randomized and treated/injected)
3-Month Evaluation | 55 | 56 | 54
6-Month Evaluation | 54 | 55 | 53
Completed | 53 | 53 | 50
Not Completed | 2 | 3 | 6
Not completed — Patient/Caregiver Preference | 2 | 2 | 3
Not completed — Death | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The efficacy/Intent-to-Treat (ITT) population comprises 167 subjects who received an intramyocardial injection of auto-CD34+ cells or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control | Total
Number analyzed (Participants) | 55 | 56 | 56 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.1) | 59.8 (9.2) | 61.8 (8.5) | 61.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 6 | 22
  Male | 46 | 49 | 50 | 145
Region of Enrollment [Number; unit: participants]
  United States | 55 | 56 | 56 | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Angina Episodes Per Week at 6 and 12 Months
Description: The number of angina episodes were collected via an electronic subject diary for four weeks at Baseline and at 6 and 12 months. The four-week angina episodes (per week mean) were used as the frequency for each visit. A lower number represents fewer angina episodes. A lower number is better.
Time Frame: 6 and 12 months
Population: Intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: angina episodes/week
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control
Number analyzed (Participants) | 50 | 50 | 46
angina episodes/week
  6 months | 6.8 (1.1) | 8.3 (1.1) | 10.9 (1.2)
  12 months | 6.3 (1.2) | 7.2 (1.1) | 11.0 (1.2)
Statistical Analysis 1: Comparison: CLBS14: Low-Dose Group vs Placebo Control; Frequency of angina episodes per week 6 months after treatment; Test type: Superiority; p = 0.020, ANCOVA
Statistical Analysis 2: Comparison: CLBS14: Low-Dose Group vs Placebo Control; Frequency of angina episodes per week 12 months after treatment; Test type: Superiority; p = 0.035, ANCOVA
Statistical Analysis 3: Comparison: CLBS14: High-Dose Group vs Placebo Control; Frequency of angina episodes per week 6 months after treatment; Test type: Superiority; p = 0.167, ANCOVA
Statistical Analysis 4: Comparison: CLBS14: High-Dose Group vs Placebo Control; Frequency of angina episodes per week 12 months after treatment; Test type: Superiority; p = 0.181, ANCOVA

2. Secondary Outcome: Exercise Treadmill Test According to Modified Bruce Protocol: Mean Change From Baseline in Duration of Exercise
Description: A modified Bruce Protocol Exercise Treadmill Test was used to evaluate duration of exercise in all subjects.
Time Frame: Change from Baseline to 6 months and change from baseline to 12 months after treatment
Population: ITT population (note that the number of participants analyzed may differ due to missing data)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control
Number analyzed (Participants) | 49 | 48 | 41
seconds
  Change from baseline to 6 months | 139 (151) | 110 (155) | 69 (122)
  Change from baseline to 12 months | 140 (171) | 103 (162) | 58 (146)
Statistical Analysis 1: Comparison: CLBS14: Low-Dose Group vs Placebo Control; Change from baseline to 6 months; Test type: Superiority; p = 0.014, ANCOVA
Statistical Analysis 2: Comparison: CLBS14: Low-Dose Group vs Placebo Control; Change from baseline to 12 months; Test type: Superiority; p = 0.017, ANCOVA
Statistical Analysis 3: Comparison: CLBS14: High-Dose Group vs Placebo Control; Change from baseline to 6 months; Test type: Superiority; p = 0.097, ANCOVA
Statistical Analysis 4: Comparison: CLBS14: High-Dose Group vs Placebo Control; Change from baseline to 12 months; Test type: Superiority; p = 0.134, ANCOVA

3. Secondary Outcome: Number of Participants With Change in Canadian Cardiovascular Society Anginal Classification Levels
Description: The Canadian Cardiovascular Society (CCS) Functional Classification of Angina is as follows:
  * Class I - Angina only during strenuous or prolonged physical activity
  * Class II - Slight limitation, with angina only during vigorous physical activity
  * Class III - Symptoms with everyday living activities, i.e., moderate limitation
  * Class IV - Inability to perform any activity without angina or angina at rest, i.e., severe limitation
Time Frame: Baseline and 12 months after treatment
Population: ITT population (note that the number of participants analyzed may differ due to missing data)
Measure: Count of Participants; unit: Participants
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control
Number analyzed (Participants) | 52 | 52 | 46
Participants
  No change in CCS classification from baseline | 16 | 19 | 16
  Improvement by 1 level (CCS) from baseline | 22 | 17 | 19
  Improvement by 2 levels (CCS) from baseline | 11 | 12 | 5
  Worsening by 1 level (CCS) from baseline | 2 | 3 | 4
  Worsening by 2 levels (CCS) from baseline | 0 | 0 | 0

4. Secondary Outcome: Changes From Baseline in Seattle Angina Questionnaire (SAQ) Scores at 6 Months
Description: Angina symptoms were evaluated based on the Seattle Angina Questionnaire (SAQ), which was used to analyze the following: physical limitations, angina stability, angina frequency, treatment satisfaction, and disease perception. The SAQ consisted of 11 questions with 5 or 6 possible responses. Responses were ordinal values (1-7, 10, 11, 97, depending on the type of question; no uniform ranges throughout); responses that corresponded to the lowest level of functioning (worse outcomes) were assigned values of 1, while responses that corresponded to higher functioning levels (better outcome) were assigned a higher ordinal value. If the response to any of these questions was 97 it was recoded as a missing value. Each scale can have a scored value ranging from 0 to 100. A larger number is better.
Time Frame: Baseline to 6 months after treatment
Population: ITT population (note that the number of participants analyzed may differ due to missing data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control
Number analyzed (Participants) | 49 | 49 | 49
score on a scale
  Physical limitations scale | 12.4 (15.6) | 10.5 (17.1) | 10.7 (15.2)
  Angina stability scale | 29.8 (30.1) | 25.5 (30.3) | 13.8 (31.9)
  Angina frequency scale | 28.3 (25.3) | 21.7 (24.6) | 26.0 (24.3)
  Treatment satisfaction scale | 11.4 (19.5) | 10.3 (21.8) | 4.9 (19.0)
  Disease perception scale | 14.4 (23.2) | 12.0 (19.4) | 15.1 (21.1)

5. Secondary Outcome: Changes From Baseline to 6 Months in Short Form 36 (SF-36) Parameters
Description: The Short Form 36 (SF-36) health survey form was used to analyze physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, general mental health, and health transition. Responses were coded as ordinal numbers going from worst (=1) to best (=highest number). These ordinal scores were transformed into scales ranging from 0 to 100. Higher numbers are generally considered better.
Time Frame: Baseline to 6 months after treatment
Population: ITT population (note that the number of participants analyzed may differ due to missing data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control
Number analyzed (Participants) | 50 | 50 | 47
score on a scale
  Physical functioning | 13.7 (18.1) | 13.2 (18.4) | 7.9 (21.8)
  Role-physical | 17.5 (35.1) | 15.9 (33.6) | 19.4 (33.2)
  Bodily pain | 13.5 (22.1) | 13.5 (21.6) | 9.4 (25.1)
  General health | 7.6 (15.5) | 6.0 (15.3) | 6.3 (15.4)
  Vitality | 14.6 (18.0) | 14.0 (20.7) | 8.9 (23.2)
  Social functioning | 16.8 (24.1) | 12.2 (24.3) | 12.0 (32.3)
  Role emotional | 10.7 (43.9) | 17.9 (51.8) | 9.7 (50.5)
  Mental health | 6.2 (16.0) | 8.4 (17.9) | 3.6 (13.6)
  Health transition | 40.4 (32.5) | 32.7 (31.1) | 29.6 (30.0)

6. Secondary Outcome: Change in Anti-anginal Medication (ie, Nitroglycerin) Use
Description: The mean nitroglycerin use per week was analyzed at baseline and 6 months
Time Frame: Baseline to 6 months
Population: ITT population (note that the number of participants analyzed may differ due to missing data)
Measure: Mean (Standard Deviation); unit: nitroglycerin use (tablets per week)
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control
Number analyzed (Participants) | 46 | 50 | 50
nitroglycerin use (tablets per week) | -6.3 (8.1) | -7.3 (9.9) | -4.2 (8.8)

ADVERSE EVENTS:
Description: The safety population comprises 174 subjects who received at least 1 dose of G-CSF.
Groups:
- No Cell or Placebo Injection: Cell mobilization with G-CSF started but no cell or placebo injection administered
Arm/Group | CLBS14: Low-Dose Group | CLBS14: High-Dose Group | Placebo Control | No Cell or Placebo Injection
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56 | 3/56 | 0/7
Serious Adverse Events (participants affected / at risk) | 21/55 | 24/56 | 32/56 | 5/7
Other Adverse Events (participants affected / at risk) | 54/55 | 52/56 | 52/56 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLBS14: Low-Dose Group (N=55) | CLBS14: High-Dose Group (N=56) | Placebo Control (N=56) | No Cell or Placebo Injection (N=7)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (3) | 1 (1) | 2 (4) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (5) | 2 (3) | 3 (4) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 8 (15) | 8 (12) | 11 (19) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (4) | 2 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (DVT) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Device lead damage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic phlebitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ischemic ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLBS14: Low-Dose Group (N=55) | CLBS14: High-Dose Group (N=56) | Placebo Control (N=56) | No Cell or Placebo Injection (N=7)
Angina Pectoris (Cardiac disorders) | 20 (25) | 14 (18) | 12 (16) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 5 (6) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (14) | 11 (16) | 9 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (6) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 5 (5) | 3 (21) | 2 (3) | 1 (1)
Fatigue (General disorders) | 15 (15) | 9 (9) | 11 (11) | 0 (0)
Edema Peripheral (General disorders) | 3 (3) | 5 (5) | 6 (6) | 0 (0)
Pain (General disorders) | 7 (8) | 9 (9) | 6 (6) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (9) | 2 (2) | 4 (5) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 14 (22) | 14 (18) | 11 (22) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (8) | 9 (9) | 4 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 6 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 12 (14) | 8 (9) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 17 (18) | 19 (25) | 11 (11) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 11 (14) | 10 (10) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (8) | 3 (4) | 5 (5) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (7) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 4 (4) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 2 (2) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 (12) | 7 (8) | 6 (7) | 0 (0)
Dizziness (Nervous system disorders) | 8 (8) | 5 (6) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 16 (20) | 25 (31) | 10 (10) | 4 (4)
Paresthesia (Nervous system disorders) | 12 (15) | 15 (15) | 17 (24) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (8) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8) | 14 (16) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 4 (5) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 6 (7) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For this study, PIs are restricted from independently publishing results before completion of a single multicenter publication or one year after study completion, whichever occurs first. Baxter requires a review of the intended publication at least 60 days prior to submission. Baxter may request an additional delay of 45 days to secure patent and/or other proprietary protection.